CLINICAL TRIAL: NCT00749788
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group Study Evaluating the Efficacy and Safety of JTT-302 Administered Daily for Four Weeks in Subjects With Low HDL-C Levels
Brief Title: Efficacy and Safety Study of JTT-302 in Subjects With Low HDL-C Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AT302-U-06-003
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): JTT-302, 200 mg
  Interventions: Drug: JTT-302
- 2 (Experimental): JTT-302, 400 mg
  Interventions: Drug: JTT-302
- 3 (Placebo Comparator): Matching placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JTT-302 — JTT-302, 100 mg tablets, 200 mg dose, oral, 30 minutes after the start of the morning meal
  Arms: 1
Drug: JTT-302 — JTT-302, 100 mg tablets, 400 mg dose, oral, 30 minutes after the start of the morning meal
  Arms: 2
Drug: Placebo — Matching placebo tablets, oral, 30 minutes after the start of the morning meal
  Arms: 3

SUMMARY:
The purpose of this study is to determine the effect of JTT-302 on the increase of High Density Lipoprotein-Cholesterol (HDL-C) levels when administered daily for four weeks in subjects with low HDL-C levels.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a Body Mass Index (BMI)≤ 35 kg/m2
* Subjects with the following lipid parameters at Visit 1 (screening visit) and Visit 3 (diet stabilization period):
* HDL-C ≤ 40 mg/dL (Men) and ≤ 50 mg/dL (Women)
* TG ≤ 500 mg/dL
* LDL-C ≤ 190 mg/dL
* Subjects who are generally healthy as determined by pre-study medical history, physical examination, vital signs and 12-lead ECG

Exclusion Criteria:

* Females who are pregnant or breast-feeding
* AST, ALT or total bilirubin ≥ 2.0 x ULN at Visit 1 (screening visit) or Visit 3 (diet stabilization period)
* Serum thyroid stimulating hormone (TSH) and levothyroxine (T4) outside of the central laboratory reference range at the screening visit
* Medical history of diabetes mellitus or two fasting serum glucose measurements > 126 mg/dL at the screening visit
* Subjects with hypertension, or two blood pressure measurements ≥ 140 mm Hg systolic or ≥ 90 mm Hg diastolic at the screening visit
* History of drug or alcohol abuse within 12 months of the screening visit
* Use of medications defined in the protocol within six-weeks prior to the screening visit and throughout the study
* Use of Cytochrome P450 3A4 inducers or inhibitors, as defined in the protocol within four weeks of the screening visit and throughout the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in HDL-C at Week 4 | 4 weeks

SECONDARY OUTCOMES:
Percent change and change from baseline at week 4 in lipid parameters | 4 weeks
Evaluate the safety profile of JTT-302 when administered for 4 weeks | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Ana, California, United States